CLINICAL TRIAL: NCT03134729
Title: PATHOS Study Pain Assessment in Thoracic Oncologic Surgery: a Prospective Randomized Trial on Pain Management After Video Assisted Major Lung Resections.
Brief Title: PATHOS Study Pain Assessment in Thoracic Oncologic Surgery
Acronym: PATHOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHT01
Record Dates: First submitted 2017-04-02; First posted 2017-05-01 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Pain, Postoperative; Lung Neoplasm
Keywords: Serratus Block, Pain Management, lung lobectomy
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized between two groups:
  Systemic analgesic therapy only (Endovenous/ Oral)
  Systemic analgesic therapy plus loco regional therapy administered under Us. guidance before the procedure (Serratus Plane Block).
  Allocation to one treatment group or another will be randomized with the aim of create two unbiased groups formed out of the same group of patients. Randomization will be provided by a software. Group allocation and treatment is overt to the investigators, but not to the patient.
Who Masked: Participant, Outcomes Assessor
Masking Description: Given the trial Design, it would be impossible to blind the caregiver about the type of treatment.
  Serratus Plan Block will be performed after the induction of General Anesthesia, the patients will thus be unaware wether being assigned to the Experimental or Control Arm.
  Clarification (May 28, 2018):
  * Nurses assess NRS (Pain Perception) and directly manage rescue doses delivery
  * Physiotherapists deliver rehab. respiratory exercises and directly assess patient's performance.
  Since their reports are directly elicited in Clinical Report Forms, they are considered outcome assessors.
  Both Nurses and Physiotherapists are unaware of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus Plane Loco-regional block (Experimental): * Continuous infusion of Tramadol 200 mg or Ketorolac 60 mg
  * Rescue analgesia with Morphine (0.1 mg/kg) a single time every 24 hours, and/or Tramadol 100 mg up to three times every 24 hours and/ or Ketorolac 30 mg up to three times every 24 hours
  plus
  Ropivacaine (30 ml, 0.3%), for Serratus Plane Block
  Interventions: Drug: Ropivacaine for Serratus Plane Block (SPB)
- Standard of Care (No Intervention): * Continuous infusion of Tramadol 200 mg or Ketorolac 60 mg
  * Rescue analgesia with Morphine (0.1 mg/kg) a single time every 24 hours and/or Tramadol 100 mg up to three times every 24 hours and/ or Ketorolac 30 mg up to three times every 24 hours

INTERVENTIONS:
Drug: Ropivacaine for Serratus Plane Block (SPB) — Serratus Plane Block (SPB) injection of low concentration Ropivacaine (30 ml, 0.3%), in the plane between the External Intercostal Muscle and the Serratus Anterior Muscle.
  Arms: Serratus Plane Loco-regional block

SUMMARY:
A randomized prospective trial to assess whether the use of loco regional anesthesia as adjuvant analgesic therapy is more effective of intravenous analgesia only.

DETAILED DESCRIPTION:
A prospective randomized trial comparing intravenous analgesia alone and in association with loco regional anesthesia consisting in a homolateral Serratus Plan Block (SPB). Loco regional blockade of the serratus is further examined by allocating the patients to two different approaches: the block being performed under US guidance by the Anesthesiologist before the beginning of the procedure, or under direct visualization, by the operating surgeon, before entering the pleural cavity.

ELIGIBILITY:
Inclusion Criteria:

* Lobectomy/ Segmentectomy plus lymphadenectomy (systematic or sampling) for cancer (not necessarily NSCLC) performed with a standardized, three portal minimally invasive approach.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Morbid obesity (BMI > 35 )
* Inability to understand and sign the Informed consent
* Proven allergy to local anesthetic drugs as required by this protocol
* Patients under chronic analgesics or neuroleptic therapy for any reason and/ or with baseline pain score (NRS scale) of 3 or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Post operative pain perception | 24 hours from the end of surgery
  Direct request to the patient to define the pain feeling, according to a Numerical Rating Scale (NRS, 0 to 10).

SECONDARY OUTCOMES:
Ability to perform post operative rehab exercises | Measured at 24 hrs and 48 hrs after surgery
  Number of forced inspiratory maneuvers during rehab respiratory exercises
Systemic rescue analgesia consumption (doses) | measured at 6 hrs, 12 hrs, 24 hrs, 36 hrs and 48hrs after surgery
  Number of extra doses of pain killers directly required by the patient (Morphine (0.1 mg/kg), Tramadol 100 mg or Ketorolac 30 mg)

CONTACTS AND LOCATIONS:
Locations (1):
- SacroCuoreDonCalabria Research Hospital, Negrar, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Result] Falcoz PE, Puyraveau M, Thomas PA, Decaluwe H, Hurtgen M, Petersen RH, Hansen H, Brunelli A; ESTS Database Committee and ESTS Minimally Invasive Interest Group. Video-assisted thoracoscopic surgery versus open lobectomy for primary non-small-cell lung cancer: a propensity-matched analysis of outcome from the European Society of Thoracic Surgeon database. Eur J Cardiothorac Surg. 2016 Feb;49(2):602-9. doi: 10.1093/ejcts/ezv154. Epub 2015 Apr 26. PMID 25913824
- [Result] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473
- [Result] Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Regional analgesia for video-assisted thoracic surgery: a systematic review. Eur J Cardiothorac Surg. 2014 Jun;45(6):959-66. doi: 10.1093/ejcts/ezt525. Epub 2013 Nov 27. PMID 24288340
- [Result] Broseta AM, Errando C, De Andres J, Diaz-Cambronero O, Ortega-Monzo J. Serratus plane block: the regional analgesia technique for thoracoscopy? Anaesthesia. 2015 Nov;70(11):1329-30. doi: 10.1111/anae.13263. No abstract available. PMID 26449303
- [Derived] Viti A, Bertoglio P, Zamperini M, Tubaro A, Menestrina N, Bonadiman S, Avesani R, Guerriero M, Terzi A. Serratus plane block for video-assisted thoracoscopic surgery major lung resection: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2020 Mar 1;30(3):366-372. doi: 10.1093/icvts/ivz289. PMID 31808538